CLINICAL TRIAL: NCT05427110
Title: Cross-sectional Study to Assess Iliotibial Band Morphometry and Stiffness Using Ultrasound Imaging in Runners With and Without Symptoms of Iliotibial Band Syndrome: a Feasibility Study
Brief Title: Shearwave Elastography in the Evaluation of Iliotibial Band Syndrome
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Nathaly Gaudreault, Researcher and Full Professor, Université de Sherbrooke
Other Study IDs: 2022-4344
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Iliotibial Band Syndrome
Keywords: Iliotibial band syndrome; Stiffness; Sonoelastography
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- asymptomatic: Runners without iliotibial band syndrome
- Iliotibial band syndrome: Runners with iliotibial band syndrome

SUMMARY:
Iliotibial band syndrome (ITBS) is a condition frequently treated in physiotherapy. The pathophysiology underlying this syndrome is still poorly understood. Ultrasound makes it possible to evaluate the morphology and to quantify, with sonoelastography (SWE), the stiffness of the iliotibial band (ITB). The objective is to determine the feasibility of a cross-sectional study aimed at evaluating the morphometry and stiffness of the ITB in runners with and without a diagnosis of ITBS. Socio-demographic and clinical data will be collected and ultrasound measurements (thickness and stiffness) of the iliotibial band will be performed in supine with the knee positioned at 2 different angles (0° and 30° flexion). Variables such as the recruitment rate/month, the inclusion/exclusion rate, the acceptability of the procedure will be used to characterize the feasibility. The relationship between ultrasound measurements and clinical outcomes will be explored. The results obtained will document feasibility issues and provide preliminary results will lay the groundwork for a large scale study.

DETAILED DESCRIPTION:
The iliotibial band (ITB) is a complex structure in which morphometry (shape, thickness, cross-sectional area) and viscoelastic properties remain poorly understood. While some hypothesize that the pain originates from friction of the ITB on the femoral condyle during knee flexion, others affirm that it is rather a compression of the ITB on the tissue underlying fat, which is highly vascularized and innervated. Current treatments in physiotherapy are based, in part, on the theory that stiffness in the ITB may contribute to iliotibial band syndrome (ITBS), resulting in prescription of stretching exercises in most rehabilitation programs. However, the plausibility of this theory remains to be demonstrated with valid and reliable instruments. Standard-mode (B-mode) ultrasound is gaining popularity for assessing ITB morphometry. However, these data remain to be correlated with the clinical symptomatology. Sonoelastography (SWE), on the other hand, is used to assess tissue stiffness. Recent studies have attempted to assess the stiffness of ITB under different experimental conditions, but these have methodological flaws (low power) and they are carried out in an asymptomatic population. This project is a first step to fill the gaps on ITB morphometry and stiffness values and explore the potential association between these factors and the clinical profile of SBIT. The primary objective is to evaluate the study the feasibility of the protocol by documenting the variables associated with this concept. Secondary objectives are: 1) To measure the stiffness of the distal BIT in runners with and without ITBS; 2) Describe the morphometry of the distal BIT in the two groups of runners; 3) Compare ITB morphometry and stiffness between the two groups of runners and 4) Investigate the association between ultrasound variables and ITBS signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 5km/week runs
* No pain during running (for healthy runners)
* For ITBS group: Received an ITBS diagnosis from a doctor or a physical therapist

Exclusion Criteria:

* Concomitant affection of the hip or knee (ex: previous fracture or surgery of the knee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All runners from Sherbrooke available during the recruitment period will be invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average of 9 months
  Proportion of included participants / total of contacts
Exclusion rate | Through study completion, an average of 9 months
  Proportion of excluded participants / total of contacts
Refusal rate | Through study completion, an average of 9 months
  Proportion of participants who refused to participate / total of contacts
Lenght of the procedure | Baseline
  Time for each evaluation in minutes
Cost of the study | Through study completion, an average of 9 months
  Cost of the patients compensation, ultrasounds gel, staff, in Canadian dollars
Acceptability of the procedure | Baseline
  opinion of participant regarding lenght of the procedure, unconfort or pain during the procedure

SECONDARY OUTCOMES:
Morphometric ITB measures | Baseline
  Thickness of distal iliotibial band with mode B ultrasound in millimeter
Stiffness of ITB | Baseline
  Stiffness of mid and distal ITB using SWE in kPa or m/s
Stiffness of TFL | Baseline
  Stiffness of TFL muscle belly using SWE in kPa or m/s
Pain intensity | Baseline
  To assess pain intensity using a Numerical Rating Scale (NRS), 0 to 10 in which 0 mean no pain and 10, the worst pain ever feeled
Knee pain and function questionnaires | Baseline
  To assess knee pain and function using the Anterior knee pain scale (AKPS). 13 questions with a total score of 100 that mean an excellent function.
Knee pain and function questionnaires | Baseline
  To assess knee pain and function using the Lower Extremity Functional Scale (LEFS) with 20 questions with a total score of 80 that mean an excellent function
Muscle retraction test | Baseline
  To assess retraction of Tensor Fascia Lata(TFL) muscle using Modified Ober Test. Score will be measure with an inclinometer in degree of the hip adduction

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly Gaudreault, Pt, Ph.D, Principal Investigator — Université de Sherbrooke
Locations (1):
- Sonia Bédard, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided